CLINICAL TRIAL: NCT03188614
Title: Different Crystalloids on the Incidence of Acute Kidney Injury in Shock Patients
Brief Title: Crystalloids for AKI in Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017ZDSYLL018P
Record Dates: First submitted 2017-03-08; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Shock
Keywords: shock; crystalloid; acute kidney injury
MeSH Terms: conditions — Shock; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline group (Placebo Comparator): Shock patients who resuscitated with normal saline were enrolled between June, 2015-June.2016.
  Interventions: Drug: Fluid resuscitation
- Balanced solution group (Experimental): Shock patients who resuscitated with balanced solution were enrolled after June, 2016.
  Interventions: Drug: Fluid resuscitation

INTERVENTIONS:
Drug: Fluid resuscitation — The placebo group is resuscitated with normal saline, the experimental group is resuscitated with balanced fluid.

SUMMARY:
Fluid resuscitation is important in shock therapy, but the choice of fluids, especially the choice of crystalloid is under debate. It is said that normal saline is related to hyperchloremia， which might lead to acute kidney injury. Thus the hypothesis of the study is to explicit whether balanced salt solution could reduce the incidence of acute kidney injury when compared with normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Shock patients

Exclusion Criteria:

* History of chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 28-day
  Diagnosis of acute kidney injury

SECONDARY OUTCOMES:
Usage of renal replacement of therapy | 28-day
  Usage of CRRT

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, Doctor, Principal Investigator — Southeast University

IPD SHARING:
Plan to Share IPD: No